CLINICAL TRIAL: NCT06487884
Title: INTRAVENOUS DRUG APPLICATIONS THROUGH ESCAPE GAMES: A MIXED METHOD RESEARCH ON THE KNOWLEDGE AND SKILL LEVELS AND LEARNING EXPERIENCES OF NURSING STUDENTS
Brief Title: INTRAVENOUS DRUG APPLICATIONS THROUGH ESCAPE GAMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ASENA KÖSE, Research Assistant, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASENA
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Nursing Students; Drug Application; Game Based Learning
Keywords: nursing students; escape games; skill; learning experience; information

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- escape games (Experimental): This group was played a 45-minute escape game.
  Interventions: Other: escape games
- control group (No Intervention): This group was not allowed to play any games other than routine nursing education.

INTERVENTIONS:
Other: escape games — A suitable day and time will be determined in the curriculum of the students in the intervention group and escape games consisting of various games involving intravenous drug administration will be played. Games will be played within the determined game guidelines. Each group will play the games at the stations respectively and get a clue at the end of each game. After completing the last game, the time it takes to find the password and complete the game will be recorded. After all groups complete the game, the group that completes the games in the shortest time will win the game and receive the prize in the chest.
  Arms: escape games

SUMMARY:
Nursing students must have sufficient competence in medication safety before starting to work in clinics. Most nursing students want to actively participate in education. Active and interesting learning activities attract more attention than lecture and instructor-oriented approaches. One of the learning methods that has attracted attention recently is the escape games technique. This study aims to determine the knowledge and skill levels and learning experiences of nursing students regarding intravenous drug administration skills using the escape games method.

DETAILED DESCRIPTION:
In global nursing education, patient safety is increasingly integrated into the nursing education curriculum based on real healthcare services. Nurses play an important role in preventing medication errors and administering safe medications. Nursing students must also have sufficient competence in medication safety before they start working in clinics. The majority of nursing students prefer to actively participate in education. Generation Z, also known as the Millennial generation, demands to participate in multi-tasking events where they receive quick responses. One of the interesting learning methods is the escape games technique. The concept of escape games is derived from recreational escape rooms. An escape room is a team game that requires a group of players to escape the room by solving a series of puzzles within a limited time. All escape room activities use a simple game loop. Games that maintain the same method but end with completing the game and reaching the reward rather than escaping from a room are called escape games. The primary aim of the research is to determine the effect of intravenous drug administration skills given through escape games on the motivation and satisfaction levels of nursing students and their views on their learning experiences. It is a mixed methods research in which quantitative and qualitative research methods are used together. The data of the research will be collected face to face from first year students studying at Atatürk University Faculty of Nursing and taking the "Principles of Nursing" course, using the "Student Information Form", "Intravenous Drug Applications Knowledge Test" and "Intravenous Drug Applications Checklist". In the qualitative part of the research, "Semi-Structured Interview Form" will be used. Quantitative data processing and statistical analysis will be done with SPSS software. Descriptive statistical methods will be used to evaluate the data, and manual coding and content analysis method will be used to analyze the qualitative data. As a result of the research, it is expected that students will be satisfied with the method used and this method will be effectively integrated into the education system.

ELIGIBILITY:
Inclusion Criteria:

Volunteering to play escape games, Being 18 years or older, Taking the Fundamentals of Nursing course for the first time, Not being a student of an exchange program such as Erasmus and having a native language of Turkish (Because these students must have sufficient command of the native language to be used in the study.) Not having received any previous training on intravenous drug administration, Not to be absent on the dates when research data will be collected.

Exclusion Criteria:

Not taking the Fundamentals of Nursing course or being exempt from the course, wanting to leave the research, not being proficient in the native language to be used in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intravenous Drug Administration Knowledge Test | 6 weeks
  This test was prepared by the researchers in line with the literature. It consists of questions regarding the achievements that students are expected to achieve within the scope of the relevant subject. The knowledge test includes 20 multiple choice questions. After these questions are created by the researchers participating in the study, they will be sent to experts in the relevant field and their opinions will be taken and their final form will be given. In terms of scope, the knowledge test created by the researchers will be sent to expert faculty members in the Department of Nursing Principles and to experts on the subject for evaluation and opinions in terms of Turkish Language. The test will be finalized in line with the recommendations from experts.
Intravenous Drug Administration Checklist | 6 weeks
  Intravenous Drug Administration Checklist consists of application steps that question the procedure steps in detail, prepared in line with the objectives of the course content. This form, prepared by the researchers, was prepared in the form of a rubric and in line with the literature in order to observe the students objectively. Intravenous Drug Administration Checklist consists of three sub-checklists titled "Application Steps of Withdrawing Medicine from Ampoule", "Application Steps of Withdrawing Medicine from Vial" and "Practice Steps of Initiating Intravenous Drug Administration"

CONTACTS AND LOCATIONS:
Locations (1):
- Asena KÖSE, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No